CLINICAL TRIAL: NCT01131832
Title: Genetic Basis for Heterogeneity in Response of Plasma Lipids to Plant Sterols
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Peter J. H. Jones, Professor, Food Science and Human Nutritional Sciences, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: B2007:073
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Hyperlipidemia
Keywords: Cholesterol, Plant sterols, Non-response, SNPs,
MeSH Terms: conditions — Hyperlipidemias | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Plant sterol (Experimental): Plant sterol supplementation, 2 grams per day of plant sterols in a margarine
  Interventions: Dietary Supplement: Plant sterol; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant sterol
Dietary Supplement: Placebo

SUMMARY:
The substantial range of individual responsiveness to plant sterols has important ramifications. Marked differences across individuals in particular aspects of the cholesterol metabolic pathway must alter the impact of plant sterol consumption. As such, a pronounced need exists to understand the genetic and metabolic factors that explain the substantial degree of heterogeneity in response of lipid concentrations to plant sterols across individuals. The primary focus of this trial is to delineate the impact of differing cholesterol synthesis levels on response of LDL-C and other plasma lipids to plant sterol consumption. Participants pre-identified as high or low endogenous cholesterol synthesizers, according to their screening level of lathosterol to cholesterol ratios, will be given PS or a placebo containing margarine to consume under supervision for 4 weeks in a crossover design. The trial will characterize the responsiveness of the participants' total, LDL, and HDL cholesterol, as well as triacylglycerol (TG) concentrations, to plant sterol consumption. This research will determine if cholesterol synthesis phenotype predicts the responsiveness of lipids to plant sterol consumption. Variations in candidate genes involved in cholesterol metabolism will also be investigated in order to find associations with both cholesterol metabolism phenotypes and responsiveness of lipids to plant sterols. The output of this research will be to advance the knowledge of which genetic factors influence the degree of cardiovascular benefit derived from plant sterols through lipid lowering.

ELIGIBILITY:
Inclusion Criteria:

* fasting serum LDL cholesterol >3.0 mmol/L
* high or low lathosterol to cholesterol ratio

Exclusion Criteria:

* smoking
* use of lipid lowering therapy
* documented cardiovascular/atherosclerotic disease
* inflammatory disease
* diabetes
* uncontrolled hypertension
* kidney disease
* liver disease
* other systemic diseases
* cancer
* chronic alcohol consumption (> 2 servings/day)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Serum Lipids | Baseline (Day 1,2) and Endpoint (Day 27,28) of each experimental period
  Total Cholesterol, LDL-C, HDL-C, Triglycerides
Serum non-cholesterol sterols | Baseline (Day 1,2) and Endpoint (Day 27,28) of each experimental period
  Lathosterol,Lanosterol,Desmosterol,Sitosterol,Campesterol,Cholestanol,
Genotype via single nucleotide polymorphism analysis | Baseline
  SNP genotyping in genes related to cholesterol metabolism

SECONDARY OUTCOMES:
Cholesterol synthesis measurement by deuterium incorporation | Endpoint (Day 27,28) of each experimental period
  Cholesterol biosynthesis will be determined as the rate of incorporation of deuterium from body water into red blood cell membrane free cholesterol over a 24 hour period (day 27 to day 28 of each period). The change in deuterium enrichment within red blood cell free cholesterol will be determined as an index of synthesis, the fractional synthesis rate (FSR) of cholesterol.
Change in cholesterol absorption due to plant sterol consumption | Change in cholesterol absorption from control period (measured over days 24-28) to plant sterol period (days 24-28)
  Ninety-six hours before the end of each period, participants will ingest 65 mg [3, 4-13C]-cholesterol. The 13C-cholesterol will be dissolved in 5 g of warmed margarine, and consumed on a slice of bread. A fasted blood sample will be taken at baseline on day 24 prior to isotope administration, as well as fasting samples on days 25, 26, 27 and 28 to monitor enrichment levels of 13C-cholesterol in plasma total cholesterol. The area under the curve of 13C-cholesterol from 0-96 hours (days 24-28) at the end of the control period will be compared to the same area under the curve at the end of the plant sterol period to determine the change in cholesterol absorption due to plant sterol consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J.H. Jones, PhD, Principal Investigator — Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Locations (2):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] MacKay DS, Eck PK, Gebauer SK, Baer DJ, Jones PJ. CYP7A1-rs3808607 and APOE isoform associate with LDL cholesterol lowering after plant sterol consumption in a randomized clinical trial. Am J Clin Nutr. 2015 Oct;102(4):951-7. doi: 10.3945/ajcn.115.109231. Epub 2015 Sep 2. PMID 26333513
- [Derived] Mackay DS, Gebauer SK, Eck PK, Baer DJ, Jones PJ. Lathosterol-to-cholesterol ratio in serum predicts cholesterol-lowering response to plant sterol consumption in a dual-center, randomized, single-blind placebo-controlled trial. Am J Clin Nutr. 2015 Mar;101(3):432-9. doi: 10.3945/ajcn.114.095356. Epub 2015 Jan 14. PMID 25733626